CLINICAL TRIAL: NCT04652128
Title: Effect of Zoledronic Acid on Prevention of Bone Loss in Acute Phase First-ever Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2019-0496
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- zoledronate (Experimental): Subject will receive a single infusion of zoledronic acid 5mg/100mL intravenously.
  Interventions: Drug: Zoledronic acid
- saline (Placebo Comparator): Subject will receive a single infusion of physiological saline 100mL intravenously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zoledronic acid — Subject will receive a single infusion of zoledronic acid 5mg/100mL intravenously.
  Arms: zoledronate
Drug: Placebo — Subject will receive a single infusion of physiological saline 100mL intravenously.
  Arms: saline

SUMMARY:
In order to reduce the incidence of fractures due to osteopenia, osteoporosis, and bone mineral density in first stroke patients, the purpose of this study was to determine whether it is meaningful to administer zoledronic acid prophylactically, and to define the characteristics of the patient group that can benefit.

Subjects suitable for the selection criteria are divided into an experimental group (zoledronic acid group) and a control group (physiological saline group) in random permuted blocks. Random assignment means that a coin is thrown and assigned to the experimental group or the control group with the probability of a head or tail, and is assigned using a random number table.

The comparison-control group was designed to analyze and compare whether there is a significant effect of preventing the decrease in bone density in the group administered zoledronic acid through the double-blind experimental group and the control group.

The reason why physiological saline was selected as a reference drug was to double-blind with zoledronic acid, because it does not affect the subject's bone density and has a very low possibility of side effects, and its transparent properties are similar to that of zoledronic acid.

Subjects undergo a bone density (BMD-Spine and femur, Whole Body Composition Assessment) test using DEXA (dual energy x-ray absorptiometry) through outpatient or hospitalization at the Department of Rehabilitation within one month after the onset of stroke.

Subsequently, the subject will receive a single infusion of zoledronic acid 5mg/100mL or physiological saline 100mL intravenously at the outpatient or inpatient ward depending on the group. Subsequently, the subject will receive a single infusion of zoledronic acid 5mg/100mL or physiological saline 100mL intravenously at the outpatient or inpatient ward depending on the group.

Each subject or guardian fills in the questionnaire form at the time of the first injection, 6 months and 12 months after the injection, and immediately sees the fractures, side effects, and changes in drugs taken from the last survey to the present.

At the first injection, 6 months and 12 months after the injection, the above examination (bone density) is performed through an outpatient department of rehabilitation medicine, and by type known to be related to zoledronic acid administration such as fractures during the period (primary fragile fracture, non-spine fragile fracture, Symptom fracture, spine fracture, etc.)

ELIGIBILITY:
Inclusion Criteria:

1. Hemiplegia due to first-ever ischemic and/or hemorrhagic stroke
2. Stroke confirmed by CT or MRI
3. Acute/Subacute stage: less than 1months after onset
4. Men or women 65 years of age or older
5. T-score between -1.0 and -2.5 (osteopenia patients)
6. Previously walk independent
7. Initial stroke severity is mild to moderately severe to very severe with an initial NIHSS score of 5 or more after the onset
8. Unable to walk 1 week after stroke onset, (Functional Ambulatory Category [FAC]<2)
9. Severe motor function involvement (Total of FMA: < 50)
10. Written informed consent

Exclusion Criteria:

1. Progressive or unstable stroke
2. Pre-existing and active major neurological disease
3. Previously diagnosed as osteoporosis
4. Lactating Mother or pregnant woman
5. Hypocalcemia(<8.8mg/dL or 2.1mmol/L), hypomagnesemia( <1.7 mg/dL or 0.7mmol/L) or Hypophosphatemia (<2.5 mg/dL or 0.81mmol/L)
6. History of Thyroid Surgery, Hypoparathyroidism or Small Intestine Excision
7. Fracture history of BMD site (L1-L5 or femur head)
8. Creatinine clearance rate <35 mL/min, Severe Renal Disease or under current treatment with an aminoglycoside antibiotic
9. Dehydration
10. Malabsorption States
11. History of Bronchial Asthma
12. Recent Invasive Dental Procedure
13. History of Aseptic Necrosis of Jaw Bone
14. A history of significant alcohol or drug abuse in the prior 3 years
15. Advanced liver, cardiac, or pulmonary disease
16. A terminal medical diagnosis consistent with survival < 1 year
17. Any Condition that would represent a contraindication to zoledronate, including allergy to zoledronate
18. Previous bisphosphonate administration history, including zoledronate

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | up to 1 month
  BMD (Spine and femur, Whole body composition assessment) test using DEXA (dual energy x-ray absorptiometry) is performed.
Bone mineral density | 6 months
  BMD (Spine and femur, Whole body composition assessment) test using DEXA (dual energy x-ray absorptiometry) is performed.
Bone mineral density | 12 months
  BMD (Spine and femur, Whole body composition assessment) test using DEXA (dual energy x-ray absorptiometry) is performed.

CONTACTS AND LOCATIONS:
Overall Officials: Deog Young Kim, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No